CLINICAL TRIAL: NCT01336179
Title: The Efficacy of the Miswak Chewing Sticks (Salvadora Persica)on Plaque Removal and Gingival Health: Randomised Clinical Trial
Brief Title: Comparative Effect of Chewing Sticks and Toothbrushing on Plaque Removal and Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Dr Tareq Abu Saleh, Department of Preventive Dental Sciences, Faculty of Dentistry, Taibah University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UTFD201127021
Record Dates: First submitted 2011-04-06; First posted 2011-04-15 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-04

CONDITIONS: Plaque Induced Gingivitis
Keywords: gingivitis; dental plaque; oral hygiene; toothbrush; chewing sticks
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Miswak, dental plaque and gingivitis (Experimental)
  Interventions: Procedure: Salvadora persica
- Toothbrush, dental plaque and gingivitis (Active Comparator)
  Interventions: Procedure: Toothbrush

INTERVENTIONS:
Procedure: Salvadora persica — twice daily use, two minutes interval
  Arms: Miswak, dental plaque and gingivitis
Procedure: Toothbrush — Twice daily use two minutes interval
  Arms: Toothbrush, dental plaque and gingivitis

SUMMARY:
The purpose of the proposed study is to compare the effect of chewing sticks (Miswak) and the toothbrushes on plaque removal and gingival health.

DETAILED DESCRIPTION:
Dental plaque removal is essential in maintaining oral health. Methods for oral hygiene vary from country to country and from culture to culture. The use of a wood stick (miswak or chewing stick) for brushing the teeth is considered an important tool for oral hygiene care in many Afro-Asian communities. The aim of the study is to compare the effect of the chewing stick (miswak), and toothbrushing on plaque removal and gingival health. The participants comprise 18 healthy Saudi Arabian male volunteers aged 21 to 30 years, at Taibah University in Saudi Arabia. The study was designed as a single, blind, randomized split-mouth study. Professional tooth cleaning was conducted, and after six weeks use of either the miswak or toothbrush on each quadrant, modified plaque and gingival indices, were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* presence of at least 14 teeth

Exclusion Criteria:

* Subjects on medications (antiinflammatory or antibiotics)

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Miswak is useful for removing plaque and preventing gingivitis | 6 weeks
  Miswak will be compared to toothbrush as a mechanical plaque control device, by calculating plaque index and gingival index scores for participants after 6 weeks of use.

CONTACTS AND LOCATIONS:
Overall Officials: Tareq AS Abu Saleh, MSc, MRD, Principal Investigator — Assistant professor in Periodontics, Taibah University
Locations (1):
- Faculty of Dentistry Taibah University, Al Madīnah, Almadinah, Saudi Arabia